CLINICAL TRIAL: NCT06244004
Title: A Randomized Open Label Phase II Trial of FDG-PET-Guided Metastasis Directed Therapy in Patients With Metastatic Hormone Sensitive Prostate Cancer: PRTY Trial: PET- Guided Radiotherapy Consolidation
Brief Title: FDG-PET-Guided Metastasis Directed Radiation Therapy for the Treatment of Metastatic Hormone Sensitive Prostate Cancer, The PRTY Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 23U09; NCI-2023-10764 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00220350; NU 23U09 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Castration-Sensitive Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Cytotoxins; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Arm 1A (FDG-PET, MDRT, SOC cytotoxic chemotherapy & ADT) (Experimental): Patients undergo an FDG-PET scan after 6 months of SOC cytotoxic chemotherapy + ADT. Patients with PET-avid disease continue their SOC ADT and undergo MDRT to up to 5 disease sites in the absence of unacceptable toxicity. Patients also undergo CT and bone scans throughout the trial.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cytotoxic Chemotherapy; Procedure: FDG-Positron Emission Tomography; Radiation: Radiation Therapy
- Arm 1B (FDG-PET, SOC cytotoxic chemotherapy & ADT) (Active Comparator): Patients undergo an FDG-PET scan after 6 months of SOC cytotoxic chemotherapy + ADT. Patients with PET-avid disease continue their SOC ADT on study. Patients also undergo CT and bone scans throughout the trial.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cytotoxic Chemotherapy; Procedure: FDG-Positron Emission Tomography
- Arm 1C (FDG-PET, SOC cytotoxic chemotherapy & ADT) (Active Comparator): Patients undergo an FDG-PET scan after 6 months of SOC cytotoxic chemotherapy + ADT. Patients without PET-avid disease continue their SOC ADT on study. Patients also undergo CT and bone scans throughout the trial.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cytotoxic Chemotherapy; Procedure: FDG-Positron Emission Tomography
- Arm 2A (FDG-PET, MDRT, SOC ADT) (Experimental): Patients undergo an FDG-PET scan after 6 months of SOC ADT. Patients with PET-avid disease continue their SOC ADT and undergo MDRT to up to 5 disease sites in the absence of unacceptable toxicity. Patients undergo an additional FDG-PET scan at 6 months. Patients also undergo CT and bone scans throughout the trial.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography; Radiation: Radiation Therapy
- Arm 2B (FDG-PET, SOC ADT) (Active Comparator): Patients undergo an FDG-PET scan after 6 months of SOC ADT. Patients with PET-avid disease continue their SOC ADT on study and undergo an additional FDG-PET scan at 6 months. Patients also undergo CT and bone scans throughout the trial.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography
- Arm 2C (FDG-PET, SOC ADT) (Active Comparator): Patients undergo an FDG-PET scan after 6 months of SOC ADT. Patients without PET-avid disease continue their SOC ADT on study and undergo an additional FDG-PET scan at 6 months. Patients also undergo CT and bone scans throughout the trial.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: FDG-Positron Emission Tomography

INTERVENTIONS:
Drug: Antiandrogen Therapy — Undergo SOC ADT
  Other Names: ADT; Androgen Deprivation Therapy; Androgen Deprivation Therapy (ADT); Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cytotoxic Chemotherapy — Receive SOC cytotoxic chemotherapy
  Other Names: Cytotoxic; Cytotoxic Therapy
  Arms: Arm 1A (FDG-PET, MDRT, SOC cytotoxic chemotherapy & ADT); Arm 1B (FDG-PET, SOC cytotoxic chemotherapy & ADT); Arm 1C (FDG-PET, SOC cytotoxic chemotherapy & ADT)
Procedure: FDG-Positron Emission Tomography — Undergo FDG-PET
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Radiation: Radiation Therapy — Undergo MDRT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm 1A (FDG-PET, MDRT, SOC cytotoxic chemotherapy & ADT); Arm 2A (FDG-PET, MDRT, SOC ADT)

SUMMARY:
This phase II trial compares the effect of FDG-positron emission tomography (PET)-guided metastasis directed radiation therapy (MDRT) in combination with standard treatments to standard treatments alone in treating patients with prostate cancer that is sensitive to androgen-deprivation therapy (ADT) and has spread from where it first started (primary site) to other places in the body (metastatic). Prostate cancer is the second leading cause of cancer death among men in the United States, despite the approval of several life-prolonging treatments by the Food and Drug Administration. However, over the past 10 years, there have been significant improvements in prolonging the lives of those with metastatic hormone sensitive prostate cancer, specifically by adding treatments to standard therapy, such as ADT. More recently, trials have demonstrated a benefit of using radiotherapy (high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors) to delay the progression of cancer and prolong life for patients with metastatic disease. Imaging scans with FDG-PET may be able to identify cancer sites that remain active despite standard treatment. Giving MDRT plus standard treatment to patients with FDG-PET-identified cancer sites may work better than standard treatment alone in treating metastatic hormone sensitive prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression free survival (PFS) between standard of care (SOC) + MDRT (Arm 1A) versus (vs) SOC alone (Arm 1B). (Cohort 1 [cytotoxic therapy cohort]) II. To compare the proportions of patients in Arm 2A vs Arm 2B who attain complete response (CR) 6 months after randomization. (Cohort 2 [non-cytotoxic therapy cohort])

SECONDARY OBJECTIVES:

I. To compare the radiographic progression-free survival (rPFS) between Arms 1A and 1B. (Cohort 1 [cytotoxic therapy cohort]) II. To determine the proportions of patients with metastatic hormone sensitive prostate cancer (mHSPC) who achieve a serum prostate-specific antigen (PSA) level < 4 ng/mL and < 0.01 ng/mL and compare them between Arm 1A and 1B. (Cohort 1 [cytotoxic therapy cohort]) III. To determine the proportion of patients with skeletal related events (SRE), and compare them between Arms 1A and 1B. (Cohort 1 [cytotoxic therapy cohort]) IV. To assess the safety and toxicity of MDRT during and following MDRT completion. (Cohort 1 [cytotoxic therapy cohort]) V. To determine the objective response rate (ORR), defined as the proportion of patients who experience a confirmed complete response (CR) or confirmed partial response (PR) on fludeoxyglucose F-18 (FDG)-PET-2, and to compare ORR between Arms 2A and 2B. (Cohort 2 [non-cytotoxic therapy cohort]) VI. To determine the progression-free survival (PFS) and radiographic progression-free survival (rPFS), and to compare between Arms 2A and 2B. (Cohort 2 [non-cytotoxic therapy cohort]) VII. To determine the proportions of patients with mHSPC who achieve a serum PSA level < 4 ng/mL and < 0.01 ng/mL (undetectable), and compare them between Arms 2A and 2B. (Cohort 2 [non-cytotoxic therapy cohort]) VIII. To determine the proportion of patients with skeletal related events (SRE), and compare them between Arms 2A and 2B. (Cohort 2 [non-cytotoxic therapy cohort]) IX. To assess the safety and toxicity of MDRT during and following MDRT completion. (Cohort 2 [non-cytotoxic therapy cohort])

EXPLORATORY OBJECTIVES:

I. To examine association between imaging features and progression free survival (Cohort 1) or likelihood of response (Cohort 2).

II. To determine the time to treatment discontinuation (TTD) in Cohort 1 Arm 1A, 1B, and 1C, and Cohort 2 Arms 2A, 2B and 2C.

OUTLINE: Patients undergoing cytotoxic chemotherapy are assigned to Cohort 1, while patients not undergoing cytotoxic chemotherapy are assigned to Cohort 2.

COHORT 1: Patients undergo an FDG-PET scan after 6 months of SOC cytotoxic chemotherapy + androgen deprivation therapy (ADT). Patients with PET-avid disease are randomized to Arm 1A or 1B. Patients without PET-avid disease are assigned to Arm 1C.

ARM 1A: Patients continue their SOC ADT and undergo MDRT to up to 5 disease sites in the absence of unacceptable toxicity. Patients also undergo computed tomography (CT) and bone scans throughout the trial.

ARM 1B: Patients continue their SOC ADT on study. Patients also undergo CT and bone scans throughout the trial.

ARM 1C: Patients continue their SOC ADT on study. Patients also undergo CT and bone scans throughout the trial.

COHORT 2: Patients undergo an FDG-PET scan after 6 months of SOC ADT. Patients with PET-avid disease are randomized to Arm 2A or 2B. Patients without PET-avid disease are assigned to Arm 2C.

ARM 2A: Patients continue their SOC ADT and undergo MDRT to up to 5 disease sites in the absence of unacceptable toxicity. Patients undergo an additional FDG-PET scan at 6 months. Patients also undergo CT and bone scans throughout the trial.

ARM 2B: Patients continue their SOC ADT on study and undergo an additional FDG-PET scan at 6 months. Patients also undergo CT and bone scans throughout the trial.

ARM 2C: Patients continue their SOC ADT on study and undergo an additional FDG-PET scan at 6 months. Patients also undergo CT and bone scans throughout the trial.

After completion of study treatment, patients are followed up at 3 months (Arms 1A, 1B, 2A, 2B only) and 6 months, and then every 6 months until 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic prostate cancer on conventional imaging (CT scan, MRI, and/or bone scan).

  * Note; Patients who had metastatic disease on conventional imaging prior to beginning ADT, but which has now resolved, are still eligible if they meet remaining eligibility criteria
* Patients must be ≥ 18 years of age at the time of informed consent.
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
* Planned treatment requirements:

  * Cohort 1

    * Patients must have mHSPC and be planning therapy with cytotoxic therapy, with or without an androgen receptor (AR) pathway inhibitor (ARPI), to be eligible for Cohort 1. Patients may also enroll if they are currently receiving or have completed cytotoxic therapy, if they are within 26 weeks +/- 4 weeks (30 weeks) of starting cytotoxic therapy and 26 weeks +/- 26 weeks (one year) of starting ADT.

      * Note:

        * Typically cytotoxic therapy means docetaxel. Patients planning other cytotoxic therapy (e.g. cabazitaxel) should discuss this with the study principal investigator (PI).
        * If a patient registers as part of cohort 1 but ends up not receiving any cytotoxic therapy, the patient may be switched to cohort 2. This must be discussed with the study PI. If the patient received at least one cycle of cytotoxic therapy, they would remain in cohort 1.
        * Patients will continue their standard of care treatment while on study (plus MDRT if they are on Arm 1A). Change in standard of care therapy will be allowed for toxicity or for de-escalation, and the patient will remain on study. Change in therapy for progression is considered a progression event.
  * Cohort 2

    * Patients must have mHSPC and be planning therapy with androgen deprivation therapy (ADT), with or without an ARPI, and not planning cytotoxic therapy, to be eligible for Cohort 2. Patients may also enroll if they are within 26 weeks +/- 4 weeks (30 weeks) of starting an AR pathway inhibitor and 26 weeks +/- 26 weeks (one year) of starting ADT.

      * Note:

        * If patients register as part of cohort 2 but end up receiving one or more cycles of cytotoxic therapy, they may be switched to cohort 1. This must be discussed with the study PI.
        * Patients will continue their standard of care treatment while on study (plus MDRT if they are on Arm 2A). If they switch therapy because of progression, they will be considered to have progressed.
        * Patients can be enrolled anytime within the initial ~6 month standard of care time period, though early enrollment is preferred. Screening can take place prior to starting standard of care (SOC) therapy or during standard of care therapy, as long as they are within 30 weeks of starting therapy.
* Leukocytes (WBC) ≥ 2,500/mcL (growth factor use allowed) (obtained prior to registration).
* Absolute neutrophil count (ANC) ≥ 1,500/mcL (growth factor use allowed) (obtained prior to registration).
* Platelets (PLT) ≥ 80,000/mcL (transfusions allowed) (obtained prior to registration).
* Patient must be able to lie flat and still for approximately 15-20 minutes AND able to tolerate FDG-PET/CT radiographical imaging and radiation treatment planning and delivery.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the endpoints for this study, in the opinion of the treating investigator, are eligible.

  * Note; Patients are ineligible if another known malignancy makes it difficult to interpret if FDG-avid lesions represent prostate cancer, or if the malignancy is expected to interfere with patients receiving standard therapy for prostate cancer for 2 years from study enrollment.
* Patients must have a life expectancy of at least 6 months, in the opinion of the treating investigator.
* Patients must have the ability to understand and the willingness to sign a written informed consent document prior to registration.

  * Note: Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.

Exclusion Criteria:

* Patients with prostate cancer that is castration resistant, which is defined as two consecutive rising PSA values despite testosterone level < 50 ng/dL.
* Patients who started androgen deprivation therapy (ADT) more than 26 weeks +/- 26 weeks (1 year) prior to enrollment.

  * Note: ADT is defined as luteinizing hormone-releasing hormone (LHRH) agonist (e.g. leuprolide, goserelin) or antagonist (e.g. degarelix, relugolix) or surgical castration. Bicalutamide 50 mg daily does not count as ADT.
  * Note: Patients will not be excluded if they were previously on intermittent therapy, as long as the current "on" period started within one year of enrollment.
* Patients who started intensification of therapy beyond ADT (e.g., AR pathway inhibitor, cytotoxic therapy) more than 26 weeks +/- 4 weeks (30 weeks) prior to registration.

  * Note: First generation antiandrogens (bicalutamide) are not considered intensification of therapy beyond ADT.
* Subjects with a known allergy to contrast material and/or contraindication to FDG-PET

  * Note: Contrast allergies: Patients with a known allergy to imaging contrast agent(s) are eligible, provided prior reactions have not been severe, and the patient is willing and able to receive pre-medications and/or supportive care according to institutional standard practice (e.g., corticosteroids, antihistamines, etc.) to manage reactions adequately.
* Patients who are enrolled in another therapeutic clinical trial that would preclude them from participating in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2027-02-18 (Estimated); Study Completion 2028-02-18 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) (Cohort 1) | From randomization to first radiographic or prostate-specific antigen (PSA)-based disease progression, or death, assessed up to 36 months
  Will be estimated using the method of Kaplan-Meier and compared between treatment arms (Arms 1A and 1B) using the log-rank test. PFS rate at 18 months following randomization will be estimated and reported with the corresponding confidence intervals.
Complete response rate (Cohort 2) | At 6 months
  Will be estimated as the proportion of patients who demonstrate response based on fludeoxyglucose F-18-positron emission tomography (FDG-PET)-2 as compared to baseline (FDG-PET-1), and will be reported with the corresponding Clopper-Pearson confidence intervals. Response rates will be compared between Arms 2A and 2B using Fisher's exact test.

SECONDARY OUTCOMES:
Radiographic PFS (rPFS) (Cohort 1) | From randomization until disease progression on computed tomography (CT) and/or bone scan, or death from any cause, assessed up to 36 months
  Will be estimated using the method of Kaplan-Meier and compared between treatment arms (Arms 1A and 1B) using the log-rank test. rPFS rate at 18 months following randomization will be estimated and reported with the corresponding confidence intervals.
Proportions of patients with metastatic hormone sensitive prostate cancer (mHSPC) who achieve a serum PSA level < 0.4 ng/mL and < 0.01 ng/mL (Cohort 1) | Up to 36 months
  Will be compared using the Fisher's exact test, and estimates by arm will be reported with the corresponding Clopper-Pearson confidence intervals.
Proportion of patients with Skeletal Related Events (SRE) (Cohort 1) | Up to 36 months
  Will be compared using the Fisher's exact test, and estimates by arm will be reported with the corresponding Clopper-Pearson confidence intervals.
Incidence of adverse events (AEs) of metastasis directed radiation therapy (MDRT) (Cohort 1) | Up to 36 months
  Will be summarized by arm using the Common Terminology Criteria in Adverse Events (CTCAE) version (v) 5.0 system organ class and term. For each subject, highest AE grade across multiple occurrences of the same event will be recorded, and the number of patients will be summarized by AE type and grade.
Objective response rate (Cohort 2) | Up to 36 months
  Defined as the proportion of patients who experience a complete response or partial response on FDG-PET-2. Will be summarized by arm and compared between Arms 2A and 2B.
PFS (Cohort 2) | From randomization to first radiographic or PSA-based disease progression, or death, assessed up to 36 months
  Will be estimated using the method of Kaplan-Meier and compared between treatment arms (Arms 2A and 2B) using the log-rank test. PFS and rate at key time points, e.g. 6 and 18 months following randomization, will be estimated and reported with the corresponding confidence intervals.
rPFS (Cohort 2) | From randomization until disease progression on CT and/or bone scan, or death from any cause, assessed up to 36 months
  Will be estimated using the method of Kaplan-Meier and compared between treatment arms (Arms 2A and 2B) using the log-rank test. rPFS at key time points, e.g. 6 and 18 months following randomization, will be estimated and reported with the corresponding confidence intervals.
Proportions of patients with mHSPC who achieve a serum PSA level < 0.4 ng/mL and < 0.01 ng/mL (Cohort 2) | Up to 36 months
  Will be summarized by arm and compared between Arms 2A and 2B.
Proportion of patients with SREs (Cohort 2) | Up to 36 months
  Will be summarized by arm and compared between Arms 2A and 2B.
Incidence of AEs of MDRT (Cohort 2) | Up to 36 months
  Will report frequency of adverse events by grade ≥ 2 assessed according to the CTCAE v 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: David VanderWeele, MD, PhD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine: Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine: Delnor, Geneva, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Northwestern Medicine: Warrenville, Warrenville, Illinois